CLINICAL TRIAL: NCT01056783
Title: A Randomized, Placebo-controlled, Double-blind, Single-centre Proof-of-concept Study of OC000459 in Adult Patients With Active Eosinophilic Esophagitis
Brief Title: Proof of Concept Study of OC000459 in Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxagen Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OC000459/013/09
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OC000459 (Experimental): OC000459 100mg twice daily
  Interventions: Drug: OC000459
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OC000459 — OC000459 100mg, twice daily, tablet
  Arms: OC000459
Drug: Placebo — Placebo tablets to match OC000459 tablets, twice daily
  Arms: Placebo

SUMMARY:
This will be a randomised, double blind, placebo controlled, parallel group evaluation of the effect of OC000459 given orally for eight weeks on active eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed and symptomatic isolated eosinophilic esophagitis.
* Relevant eosinophil tissue inflammation as demonstrated by a mean eosinophil load >= 20 eos/hpf in 8 biopsies at the baseline visit.
* Able to swallow placebo medication successfully under supervision in the clinic
* Free of all medications for EoE (including topical steroids) for at least 2 weeks prior to baseline and free of systemic steroids for at least 90 days before screening. A proton-pump inhibitor is allowed if required for treatment of secondary acid reflux.

Exclusion Criteria:

* Other causes of esophagitis (GERD, peptic ulceration, infection etc.)
* Other causes of eosphagaeal or generalized eosinophilia (i.e. hypereosinophilic syndromes, parasitic infection, GERD)
* The patient's EoE is dependant on the level of seasonal allergens and the patient's participation in the study will occur during the allergy season.
* History of abnormal gastric or duodenal eosinophilia (e.g. HES, Churg Strauss vasculitis, EG or a parasitic infection)
* Receipt of forbidden prescribed or over the counter medication within the 4 weeks prior to the baseline visit and for the duration of the trial, including vitamins and herbal remedies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Effect of OC000459 on eosinophil load of the esophageal tissue | 8 weeks

SECONDARY OUTCOMES:
Effect of OC000459 on clinical manifestations of EoE | 8 weeks
Effect of OC000459 on endoscopic alterations | 8 weeks
Effect of OC000459 on EoE related blood and tissue biomarkers | 8 weeks
Safety and tolerability of OC000459 in patients with active EoE | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alex Straumann, Dr, Principal Investigator — Swiss EoE Research Group
Locations (1):
- Swiss EoE Research Group, Olten, Switzerland